CLINICAL TRIAL: NCT02346851
Title: The Effects of Accelerometer Triggered Functional Electrical Stimulation on Post-Stroke Hemiplegic Shoulder Subluxation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2012-0602
Record Dates: First submitted 2015-01-15; First posted 2015-01-27 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Post-Stroke Hemiplegic Shoulder Subluxation
MeSH Terms: interventions — proto-oncogene protein c-fes-fps; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- triggered FES (Experimental)
  Interventions: Procedure: Functional Electrical Stimulation (FES) treatment
- conventional FES (Active Comparator)
  Interventions: Procedure: Functional Electrical Stimulation (FES) treatment
- control group (No Intervention)

INTERVENTIONS:
Procedure: Functional Electrical Stimulation (FES) treatment — This study is randomized controlled trial performed by Random permuted blocks. This study has 2 experimental groups and 1 control group. Both experimental group receive FES treatment of their posterior deltoid and supraspinatus. Experimental group 1(Acceleration group) uses Novastim CU FS1 once a day for 30 minutes during 3 weeks. During treatment patient give a maximal effort for shoulder abduction. Experimental group 2 (Convention group) receive cyclic FES treatment for reducing shoulder subluxation. All patients have evaluation pre-intervention, post-intervention, 3 weeks after intervention and 9 weeks after intervention including physical examination and x-ray.
  Arms: conventional FES; triggered FES

SUMMARY:
Post stroke hemiplegia patient have shoulder subluxation in affected side. The investigators use functional electrical stimulation in posterior deltoid and supraspinatus for prevention and treatment. But the investigators hypothesis self triggered myoelectric stimulation system has more effective for shoulder subluxation. The purpose of this study is to compare post-stroke shoulder subluxation treatment FES and triggered FES.

ELIGIBILITY:
Inclusion Criteria:

1. Within 3months after stroke
2. 1st stroke patients with hemiplegic shoulder subluxation which is measured above one finger breadth by physical examination
3. Shoulder abduction strength is above P- grade (MMT)
4. Male or female, ≥ 20 years of age
5. Written informed consent has beed obtained
6. Patients who understand purpose of this study and conform with intervention process

Exclusion Criteria:

1. Quadriplegia or double hemiplegia
2. History of injury, surgery, etc. of U/E and upper chest area
3. person who implanted metalic device(ex. pacemaker, vagus nerve stimulator)
4. patients who have lower motor neuron lesion
5. person who have difficulty using electrode due to skin problem such as skin ulcer or open wound
6. who have seizure or epilepsy history
7. Female who are pregnant

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2013-11-12; Primary Completion 2015-09-16 (Actual); Study Completion 2015-09-16 (Actual)

PRIMARY OUTCOMES:
Difference of vertical distance | 12 weeks

SECONDARY OUTCOMES:
Physical examination of affected side | 12 weeks
Difference of joint distance of shoulder A-P radiograph | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Severance hospital, Seoul, South Korea

REFERENCES:
- [Background] Ikai T, Tei K, Yoshida K, Miyano S, Yonemoto K. Evaluation and treatment of shoulder subluxation in hemiplegia: relationship between subluxation and pain. Am J Phys Med Rehabil. 1998 Sep-Oct;77(5):421-6. doi: 10.1097/00002060-199809000-00012. PMID 9798835
- [Background] Chaco J, Wolf E. Subluxation of the glenohumeral joint in hemiplegia. Am J Phys Med. 1971 Jun;50(3):139-43. No abstract available. PMID 5579071
- [Background] Chan MK, Tong RK, Chung KY. Bilateral upper limb training with functional electric stimulation in patients with chronic stroke. Neurorehabil Neural Repair. 2009 May;23(4):357-65. doi: 10.1177/1545968308326428. Epub 2008 Dec 12. PMID 19074684
- [Background] Embrey DG, Holtz SL, Alon G, Brandsma BA, McCoy SW. Functional electrical stimulation to dorsiflexors and plantar flexors during gait to improve walking in adults with chronic hemiplegia. Arch Phys Med Rehabil. 2010 May;91(5):687-96. doi: 10.1016/j.apmr.2009.12.024. PMID 20434604
- [Background] Tong KY, Mak AF, Ip WY. Command control for functional electrical stimulation hand grasp systems using miniature accelerometers and gyroscopes. Med Biol Eng Comput. 2003 Nov;41(6):710-7. doi: 10.1007/BF02349979. PMID 14686597
- [Background] Lau H, Tong K. The reliability of using accelerometer and gyroscope for gait event identification on persons with dropped foot. Gait Posture. 2008 Feb;27(2):248-57. doi: 10.1016/j.gaitpost.2007.03.018. Epub 2007 May 21. PMID 17513111
- [Background] Koyuncu E, Nakipoglu-Yuzer GF, Dogan A, Ozgirgin N. The effectiveness of functional electrical stimulation for the treatment of shoulder subluxation and shoulder pain in hemiplegic patients: A randomized controlled trial. Disabil Rehabil. 2010;32(7):560-6. doi: 10.3109/09638280903183811. PMID 20136474